CLINICAL TRIAL: NCT00892359
Title: The Pharmacokinetics of Anidulafungin During Continuous Venovenous Hemofiltration
Brief Title: Anidulafungin During Continuous Venovenous Hemofiltration (CVVHF)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Florian Thalhammer, M.D., Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.1 - Leitner
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-04

CONDITIONS: Acute Renal Failure; Infection
Keywords: pharmacokinetics; renal replacement therapy; hemofiltration; anidulafungin
MeSH Terms: conditions — Acute Kidney Injury; Infections | interventions — Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anidulafungin (Experimental)
  Interventions: Drug: Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin — treatment for 3 days, 200 mg intravenously on the first treatment day and 100 mg on the 2 following treatment days each.

SUMMARY:
The purpose of this trial is to study the pharmacokinetics of anidulafungin during continuous venovenous hemofiltration.

Background: Anidulafungin is a cyclic lipopeptide antifungal agent of the echinocandin class. Members of this class of antifungal agents are known to inhibit the synthesis of glucan polymers in fungal cell walls. The spectrum of activity of anidulafungin includes Candida (all species, including strains resistant to fluconazole), Aspergillus, and Pneumocystis.

In intensive care patients continuous venovenous haemodiafiltration (CVVHF) is a well-established extracorporal renal replacement therapy with a high clearance rate.

Pharmacokinetic studies of antifungal agents in critically ill patients treated with CVVHF are rare. No data about anidulafungin in CVVHF are available although intensive care patients are perfect candidates for anidulafungin treatment due to their high risk profile for systemic fungal infections.

Study objective: The study is conducted to investigate the pharmacokinetics of anidulafungin during CVVHF in critically ill patients.

Study design: open, 1 arm

Study population: 10 critically ill adult patients administered to the ICU with acute renal failure and suspected or proven fungal infection.

Treatment/Dosage/Route: On the first day 200 mg of anidulafungin will be administered intravenously over 3 hours (loading dose). The following days 100 mg of anidulafungin will be administered intravenously over 1.5 hours.

Main outcome variables: The following pharmacokinetic parameters will be determined: area under the curve (AUC), half-live (t1/2), maximum plasma concentration (Cmax) and elimination fraction.

Methods: High pressure liquid chromatography (HPLC) will be used to determine anidulafungin concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 70 years
* Suspected or proven infection requiring parenteral antifungal therapy.
* Continuous venovenous hemofiltration because of an acute renal failure.

Exclusion Criteria:

* Known history of hypersensitivity to echinocandins.
* An expected survival of less than three days.
* Known alcohol dependency, epilepsy, pregnancy or liver failure.
* Neutropenic patients

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Anidulafungin area under the curve (AUC), half-live (t1/2), maximum plasma concentration (Cmax) and elimination fraction. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria